CLINICAL TRIAL: NCT06867510
Title: Preoperative Ultrasound-Guided Intermediate Cervical Plexus Block Versus Preoperative Cervical Erector Spinae Plane Block for Anterior Cervical Spine Surgery: A Randomized Controlled Study
Brief Title: Preoperative Block for Anterior Cervical Spine Surgery
Acronym: ESPB/ICPB
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Abd Elfatah khodair, Assistant lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Block in Spine Surgery
Record Dates: First submitted 2025-02-21; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Anesthesia, Local
Keywords: Regional anesthesia in cervical spine surgery
MeSH Terms: interventions — Dental Occlusion; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: All blocks will be conducted under sterile conditions in the operating room with sedation "midazolam 0.03-0.05 mg/kg as needed" 30 minutes before induction of general anesthesia.
  a total volume of 15 ml of 0.25% bupivacaine will be injected bilaterally. The spread of the local anesthetic will be visualized using ultrasound guidance. The same steps will be repeated on the other side
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intermediate cervical plexus block (Active Comparator): The patient will be positioned supine with a slight elevation of the head and the head turned away from the blocked side. After sterilizing the skin, the ultrasound probe will be placed over the middle of the posterior border of the sternocleidomastoid muscle. The needle will be inserted in-plane while keeping the probe in a transverse position. The needle tip will be placed under the sternocleidomastoid muscle and below the superficial fascia, and then, a total volume of 15 ml of 0.25% bupivacaine will be injected bilaterally. The spread of the local anesthetic will be visualized using ultrasound guidance. The same steps will be repeated on the other side.
  Interventions: Procedure: Block for Anterior Cervical Spine Surgery
- Cervical Erector spinae block (Active Comparator): The patient will be positioned laterally, with a pillow under their head. Transverse ultrasound scanning of the lower cervical area will be done. Starting from the supraclavicular brachial plexus, the transducer will be slid in a cephalic direction to show the transverse process of the C7 vertebra. Then, it will be moved further cephalic to display the transverse process of C6, along with its characteristic anterior and posterior tubercles. The transducer will be then slid posteriorly to show the posterior tubercle of C6, along with the posterior neck muscles above it (trapezius, levator scapula, and erector spinae). After prepping and draping the patient using aseptic technique, the needle will be inserted (in plane technique from posterior) until it will reach the posterior tubercle of C6. Then, a total volume of 15 ml of bupivacaine 0.25% will be injected bilaterally. The same steps will be repeated on the opposite side.
  Interventions: Procedure: Block for Anterior Cervical Spine Surgery
- Control group (Placebo Comparator): Total volume of 15 ml of saline 0.9% will be injected subcutaneous bilaterally
  Interventions: Drug: Saline (NaCl 0,9 %) (placebo)

INTERVENTIONS:
Procedure: Block for Anterior Cervical Spine Surgery — The patient will be positioned supine with a slight elevation of the head and the head turned away from the blocked side. After sterilizing the skin, the ultrasound probe will be placed over the middle of the posterior border of the sternocleidomastoid muscle. The needle will be inserted in-plane while keeping the probe in a transverse position. The needle tip will be placed under the sternocleidomastoid muscle and below the superficial fascia, and then, a total volume of 15 ml of 0.25% bupivacaine will be injected bilaterally. The spread of the local anesthetic will be visualized using ultrasound guidance. The same steps will be repeated on the other side
  Arms: Cervical Erector spinae block; Intermediate cervical plexus block
Drug: Saline (NaCl 0,9 %) (placebo) — Total volume of 15 ml of saline 0.9% will be injected subcutaneous bilaterally
  Arms: Control group

SUMMARY:
The purpose of this clinical trial study is to compare the analgesic effects of ultrasound-guided intermediate cervical plexus block Versus cervical erector spinae block in patients undergoing anterior cervical spine surgery.

* The main questions it aims to answer are:

  * The primary outcome will be recording postoperative pain intensity using Numerical Rating Scale (NRS).
  * The secondary outcomes will be measuring the performance time, onset of the sensory block, intraoperative fentanyl consumption, time to the first call for rescue analgesia (nalbuphine), postoperative total nalbuphine consumption, and postoperative complications such as nausea, vomiting, hypotension, and bradycardia.
* We will compare two blocks to a placebo.
* Participants will:

  * undergo ultrasound-guided intermediate cervical plexus block or cervical erector spinae block or a placebo
  * Be assessed for pain after 2 h, 4 h, 6 h, 12 h, and 24 h postoperatively

DETAILED DESCRIPTION:
Anterior cervical spine surgery is a common procedure for treating disc herniation, spinal cord vascular diseases, cervical spondylosis, and tumors. Cervical spine surgery is one of the most painful surgical operations, ranked among the 6 most painful out of 179 assessed surgical procedures, underscoring the challenges in pain management for this patients. Many patients requiring spine surgery are also overweight, have substance use disorders and other comorbidities related to aging.

Surgeons have been able to effectively treat patients with various cervical spine conditions by using specialized retractors, natural muscle planes, and paying careful attention to surrounding structures. However, despite the high success rates associated with these surgeries, patients often experience postoperative pain between the shoulder blades and in the neck.

Improper perioperative pain management after anterior cervical spine surgery can impact a patient's recovery, overall health, ability to swallow, may lead to nausea, vomiting, and chronic pain. Thus, effective pain management techniques are crucial to enhance postoperative care for these patients.

A regional analgesia block is a technique used to suppress nerve transmission and alleviate or prevent pain. It is commonly used in combination with general anesthesia or as the sole anesthetic technique, particularly in plastic, orthopedic and vascular surgeries to reduce the amount of anesthetic and analgesic agents needed, minimize systemic side effects, improve recovery, provide better postoperative pain relief, and shorten hospital stays.

The cervical plexus is made up of the ventral rami of the C1-C4 spinal nerves. The cervical plexus consists of motor (phrenic nerve, direct muscle branches) and terminal sensory branches (C2-C4): the supraclavicular nerves, the lesser occipital nerve, greater auricular nerve, and transverse cervical nerve. The latter is formed in the compartment between the prevertebral and superficial layer of the cervical fascia, deep to the sternocleidomastoid. Before 2004, any cervical plexus blocks that were performed superficially to the prevertebral fascia were termed superficial cervical plexus blocks. However, Telford and Stoneham suggested the term intermediate cervical plexus block to distinguish between the superficial block (subcutaneous or subplatysmal) and the block in the interfascial compartment. Intermediate cervical plexus block is a safe, popular, easy, and effective technique for regional analgesia of cervical region. The use of ultrasound guidance reduces the risk of complications, allows for real-time visualization of anatomical structures, and helps guide needle placement.

Bilateral cervical erector spinae block using ultrasound has recently been studied for shoulder surgery. Since the brachial plexus, phrenic nerves, cervical nerve roots, and deep cervical muscles are enclosed in the prevertebral fascia, injecting a local anesthetic near the cervical transverse process can spread to nearby structures within the prevertebral compartment. In a cadaver study, it was found that injecting a 20 mL dye solution into the transverse process of C6 or C7 resulted in staining of the C5-T1 nerve roots.

With the increasing number of nerve block techniques available, anesthesiologists may have difficulty determining the most appropriate technique to achieve optimal recovery after anterior cervical spine surgery. Therefore, this study will conducted to compare the efficacy of ultrasound-guided intermediate cervical plexus block and cervical erector spinae block in patients undergoing anterior cervical spine surgery.

ELIGIBILITY:
Inclusion Criteria:

* Both sex
* Age: between 21 and 60 years
* Physical status: belongs to American Society of Anesthesiologists (ASA) I, II
* Body mass index (BMI): from 25 to 30 kg/m2
* Type of surgery: elective anterior cervical spine surgery under general anesthesia

Exclusion Criteria:

* Refusal of participation.
* local infection at the puncture site.
* Mental or physical disability.
* History of allergy to study drugs (bupivacaine, fentanyl).
* Hematological disorders including coagulation abnormalities.
* Severe hepatic or kidney impairment.
* Chronic pain.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
change in postoperative pain intensity using Numerical Rating Scale | (Day 1) 30 minutes, 2 hours, 4 hours, 6 hours, 12 hours, and 24 hours postoperative
  Numeric Rating Scale ( NRS) score, a commonly used 11-point numeric scale ranges from '0' representing one pain extreme (no pain) to '10' representing the other pain extreme ( pain as bad as you can imagine or worst pain imaginable). The patient will be instructed to mark along the line to represent the intensity of pain currently being experienced.

SECONDARY OUTCOMES:
Change in the time of performance of the technique in minutes. | Perioperative/Periprocedural
  Time of performance of the technique: the time from probe insertion until the visualization of local anesthetic spread in minutes.
Change in the time to the first call for analgesia (nalbuphine) in hours. | Perioperative/Periprocedural
  The time to the first call for rescue analgesia (nalbuphine), which is the time between the end of surgery and the first report of postoperative pain, will be recorded in hours.
The total measure of nalbuphine given to each patient during the first 24 hours of the postoperative period | Perioperative/Periprocedural
  The total amount of nalbuphine in milligrams given to each patient during the first 24 hours of the postoperative period will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Teaching Hospital, Tanta, Qism Awwal Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kamel AAF, Fahmy AM, Fathi HM, Elmesallamy WAEA, Khalifa OYA. Regional analgesia using ultrasound-guided intermediate cervical plexus block versus cervical erector spinae block for anterior cervical spine surgery: a randomized trial. BMC Anesthesiol. 2024 Apr 22;24(1):153. doi: 10.1186/s12871-024-02533-6. PMID 38649826
- [Result] Abdelhaleem NF, Youssef EM, Hegab AS. Analgesic efficacy of inter-semispinal fascial plane block in Patients undergoing Cervical Spine Surgery through Posterior Approach: a randomized controlled trial. Anaesth Crit Care Pain Med. 2023 Aug;42(4):101213. doi: 10.1016/j.accpm.2023.101213. Epub 2023 Mar 7. PMID 36894055
- See also: Related Info — https://doi.org/10.1186/s12871-024-02533-6